CLINICAL TRIAL: NCT05439551
Title: A Prospective Multi-center Sample Collection Study for Evaluating the Analytical Equivalency of Serum and Whole Blood Samples Run on the MeMed Key® Platform ("Perseverance" Study)
Brief Title: Evaluating the Analytical Equivalency of Serum and Whole Blood Samples Run on the MeMed Key® Platform (Perseverance Study)
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MMD012WB
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2022-06

CONDITIONS: Acute Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pediatric and adults suspected of acute bacterial or viral infection: ED, Hospital admitted, and urgent care center patients over the age of 90 days, with clinical suspicion of acute bacterial or viral infection.
  Interventions: Diagnostic Test: MeMed BV®

INTERVENTIONS:
Diagnostic Test: MeMed BV® — Patients Serum and Whole blood samples will be examined using the MeMed BV® test. Test results will have no impact on patient management.

SUMMARY:
This is a Prospective, multi-center, sample collection study enrolling pediatric and adult subjects presented to the ED/Urgent care, with symptoms consistent with acute bacterial or viral infection will be recruited according to eligibility criteria. The study is designed to measure the MeMed BV®️ score in whole blood and serum samples and demonstrate the equivalence between the two matrices. Patients will be managed according to the current standard of care per standard institutional procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from the patient or his/her legal guardian. For children under 18 years old, written informed consent from the legal guardian must be obtained and assent from the patient may be required depending on the local requirements.
2. Over 90 days of age.
3. Clinical suspicion of acute bacterial or viral infection.
4. Symptoms of acute infectious disease < 7 days.
5. Experienced fever at least once within the last 7 days (self-reported or Temperature ≥ 37.8°C (100°F)).

Exclusion Criteria:

1. HIV, HBV, active HCV, or active Tuberculosis infection (self-declared or known from medical records).
2. Suspicion and/or confirmed diagnosis of infectious gastroenteritis/ colitis.
3. Active inflammatory disease (e.g., IBD, SLE, JIA, RA, Kawasaki, other vasculitis).
4. Pregnancy- self reported or medically confirmed.
5. Active malignancy.
6. Congenital or acquired immune deficiency (CID).
7. A proven or suspected infection on presentation with Mycobacterial (e.g., Tuberculosis, MAC), parasitic or fungal (e.g., Candida, Histoplasma, Aspergillus) pathogen.
8. Significant trauma or burns in the last 7 days.
9. Patients that have undergone major surgery in the last 7 days.
10. Current treatment with immune-suppressive or immune-modulating therapies, including without limitations:

    1. Administration of P.O.\IV\IM high dose steroids >1mg/kg/day prednisone (or equivalent) at some point in the past 10 days or daily continuous use of steroids > 0.25 mg/kg/day in the past 7 days
    2. Monoclonal antibodies, anti-TNF agents
    3. Intravenous immunoglobulin (IVIG)
    4. Cyclosporine, Cyclophosphamide, Tacrolimus, Azathioprine, Methotrexate
    5. G/GM-CSF, Interferons.

Min Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ED, Hospital admitted, and urgent care center patients over the age of 90 days, with clinical suspicion of acute bacterial or viral infection.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Measuring the MeMed BV® score with whole blood and serum samples from patients suspected of acute bacterial or viral infection and demonstrating the equivalence between the two matrices. | Through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Maimonides Medical Center, Brooklyn, New York
  - Urgent Care Clinical Trials @ AFC Urgent Care- Easley, Easley, South Carolina
- Israel (3):
  - Hillel Yaffe Medical Center, Hadera
  - Carmel Medical Center, Haifa
  - Sourasky Medical Center - Ichilov, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes